CLINICAL TRIAL: NCT07176663
Title: Safety and Effectiveness of Tirzepatide(Spartina )in Chronic Kidney Failure a Single-center Study
Brief Title: Efficacy and Safety of Tirzepatide (Spartina) in Chronic Kidney Failure
Acronym: Tirzepatide
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Associate Professor of Nephrology, Shahid Beheshti University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBMU-1404-06
Record Dates: First submitted 2025-09-05; First posted 2025-09-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spartina (Experimental): weekly injection of Tirzepatide (Spartina)
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — 2.5 mg weekly first month and 5 mg weekly for two month
  Other Names: Spartina

SUMMARY:
Diabetes management presents a complex clinical scenario marked by several challenges, especially in chronic kidney failure. These include navigating potential drug interactions between oral antidiabetic therapies and other agents. Furthermore, these patients may experience various adverse drug effects, such as lactic acidosis, electrolyte abnormalities such as hypomagnesemia, fluid retention, and lipid derangements, which can further augment overall morbidity. Consequently, many patients receive insulin. However, prolonged intensive insulin therapy may be linked to several adverse outcomes, including an increased risk of hypoglycemia and weight gain.

Hence, a common practice is to transition to medications commonly used other populations of patients. With their established benefits on glycemic control, cardiovascular health, renal benefits, and weight management, in conjunction with the aforementioned adverse effects associated with other oral antidiabetics agents, glucagon-like peptide-1 receptor agonists have emerged as an attractive therapeutic option for patients with kidney failure.

DETAILED DESCRIPTION:
Investigators will conduct a single-center clinical trial at Labafinezhad Hospital in Tehran, Iran. Initially, 15 stable chronic kidney failure patients with a glomerular filtration rate < 30 cc/min but not on dialysis, will receive tirzepatide(Spartina) therapy. Inclusion criteria consisted of age ≥18 years and a history of chronic kidney failure with preexisting diabetes or obesity with a body mass index over 27.

. Major exclusion criteria included similar drug therapy for a duration of less than 3 months and nonadherence to tirzepatide therapy. After an initial screen, investigators will enroll 15 patients who meet the inclusion criteria. The project is pending Institutional Research Ethics Committee of Shahid Beheshti University of Medical Sciences approval.

Data collection at baseline involves gathering demographic information, including age, sex, weight, height, and blood type group. Furthermore, investigators will obtain information related to past medical history, including the presence of preexisting diabetes mellitus, the onset of diabetes mellitus, and the requirement of insulin therapy. Efficacy endpoints include alterations in weight, body mass index (in kilograms divided by height in meters squared), serum triglycerides, insulin requirements, fasting plasma glucose, and estimated glomerular filtration rate, computed based on the Chronic Kidney Disease Epidemiology 2021 collaboration formula. For safety outcomes, investigators will review serum lipase, thyroid-stimulating hormone levels, and liver function tests at baseline and after tirzepatide therapy. Investigators will also report on all-cause mortality. Efficacy and safety endpoint data will be collected initially at baseline (therapy initiation) and at the end of 1 and 3d months.

ELIGIBILITY:
Inclusion Criteria:

age ≥18 years and history of diabetes or BMI over 27

Exclusion Criteria:

Previous usage of similar therapy for less than 3 months owing to the inability to capture all efficacy and safety endpoints within this brief timeframe and/or nonadherence to tirzepatide therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
weight loss | kilogram of weight loss measured by same scale one and three month after injection

CONTACTS AND LOCATIONS:
Overall Officials: Nooshin Dalili, MD, Principal Investigator — SBMU
Locations (1):
- Nooshin Dalili, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No